CLINICAL TRIAL: NCT06851494
Title: Safety and Efficacy of Linnea Safe PMMA 30% Use for Gluteal Augmentation.
Acronym: LinneaSafe30
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LEBON PRODUTOS QUIMICOS E FARMACEUTICOS LTDA. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LEBON_01_2025
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Gluteal Augmentation
Keywords: buttock augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PMMA (Experimental): Gluteal Augmentation with Linnea Safe (PMMA).
  Interventions: Device: PMMA

INTERVENTIONS:
Device: PMMA — Safety and efficacy evaluation of PMMA LinneaSafe 30% use for gluteal augmentation. Linnea Safe is a water-based gel containing Polymethylmethacrylate (PMMA) in concentrations of 2%, 10% or 30%. LInnea Safe is indicated for facial and body volumetric correction in cases of lipodystrophy due to the use of antiretrovirals in HIV-positive patients. It is also indicated for facial volumetric correction, and can be used in nasolabial folds, glabellar lines, corners of the mouth, upper lip lines, chin lines/chin lines, in the malar region, in acne scars, on the nose, to increase lips and facial contour.

SUMMARY:
This pre-market, interventional, single-arm study aims to evaluate the safety and efficacy of LinneaSafe 30% polymethylmethacrylate (PMMA) for gluteal augmentation. The study will include 119 patients, with a total recruitment of 137 to account for a 15% drop-out rate. Eligible participants are men and women over 18 years old who express interest and are deemed suitable for the procedure. The primary safety outcome is the incidence of adverse events, while the primary efficacy outcome is patient satisfaction.

DETAILED DESCRIPTION:
This pre-market, interventional, single-arm study aims to evaluate the safety and efficacy of LinneaSafe 30% polymethylmethacrylate (PMMA) for gluteal augmentation. The study will include 119 patients, with a total recruitment of 137 to account for a 15% drop-out rate. Eligible participants are men and women over 18 years old who express interest and are deemed suitable for the procedure. The primary safety outcome is the incidence of adverse events, while the primary efficacy outcome is patient satisfaction.

Patient recruitment will be conducted via social media. After signing the consent form, participants will undergo screening, including laboratory tests, gluteal ultrasound, and bioimpedance. The procedure (T0) involves baseline photos, gluteal measurements, and intramuscular PMMA augmentation (maximum 300 mL), followed by an evaluation of patient and clinician satisfaction. Follow-ups include online assessments at T1 week and T3 months to monitor adverse events. At T6 months, patients will undergo clinical evaluation, laboratory tests, photos, and satisfaction assessments, with the possibility of a retouch (up to 120 mL) if necessary, followed by an additional online check-up after one week. The final evaluation at T12 months will include photos, gluteal measurements, laboratory tests, ultrasound, bioimpedance, and an overall assessment of safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women;
* Older than 18 years;
* Signed Informed Consent Form;

Exclusion Criteria:

* Prior intramuscular filling with PMMA for volumization of the buttocks or other body areas (reported by the patient or verified on ultrasound).
* Clinical history or evidence on ultrasound of intramuscular injection of liquid/industrial silicone, hydrogels (except hyaluronic acid and absorbable biostimulators performed up to 6 months before), synthol, potenay, ADE vitamins or other products in the glutes
* Pregnant or breastfeeding women
* Presence of silicone prosthesis for gluteal augmentation;
* Levels of 25 hydroxy vitamin D > 60 mg/mL;
* Vitamin D supplementation in the 3 months prior to the procedure - even with 25 hydroxy vitamin D levels between 15 and 60 mg/mL
* Altered PTH (less than 12pg/mL or greater than 65 pg/mL CRP greater than 1 mg/dL (or 10 mg/L)
* Erythrocyte sedimentation value 2 times higher than normal;
* Women with testosterone levels greater than 70 ng/dL
* Women with estrogen levels greater than 450 pg/mL
* Urea value greater than 50 mg/dL
* Creatinine value greater than 1.3 mg/dL
* Glomerular filtration rate less than 90 mL/min
* Rheumatoid factor value greater than 79 UI/mL
* Ionic calcium values greater than 5.2 mg/dL (or 1.30 mmol/L)
* Total calcium value greater than 10.5 mg/dL
* Iron value greater than 175 µg/dL
* Ferritin value greater than 336 ng/dL
* Calcitriol greater than 90.1pg/dL
* Uncontrolled diabetes (fasting blood glucose > 100mg/dL)
* Antinuclear factor (ANA) > 1:160;
* Personal history of more than one episode of pain due to kidney stones (except during pregnancy)
* Ratio of urinary calcium and urinary creatinine in an isolated urine sample > 250.
* Patients using medications for cancer treatment
* Patients with lupus, systemic scleroderma, dermatomyositis, granulomatous diseases
* Any other contraindications mentioned in the product's instructions for use, such as: history of evolving autoimmune disease, during treatment with immunosuppressants, or in any disorder or active skin infection. The use is absolutely contraindicated in cases of active herpes lesions. In cases of herpetic history, prophylactic treatment is recommended. Any inflammatory reaction from injections is also a contraindication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | From enrollment to the end of treatment at 12 months
  Expected events will be classified as adverse events when they persist for more than two weeks, and must be reported throughout the study. Adverse events not previously identified will also be monitored at all visits.

SECONDARY OUTCOMES:
Patient Satisfaction | From enrollment to the end of treatment at 12 months
  Patient and physician satisfaction will be evaluated using the Portuguese version of the Global Aesthetic Improvement Scale, assigning values according to the following parameters:
  Very much improved (5): excellent cosmetic result after the procedure. Much improved (4): marked improvement in the appearance of the initial condition, but not completely optimal for the patient.
  Improved (3): obvious improvement in the appearance of the initial condition. No change (2): appearance is essentially the same as the original condition. Worse (1): appearance is worse than the original condition. The satisfaction assessment will be conducted at the T6 and T12 visits.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Bortolozo, Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lemperle G, Morhenn V, Charrier U. Human histology and persistence of various injectable filler substances for soft tissue augmentation. Aesthetic Plast Surg. 2003 Sep-Oct;27(5):354-66; discussion 367. doi: 10.1007/s00266-003-3022-1. Epub 2003 Dec 4. PMID 14648064
- [Background] Chacur R, Sampaio Menezes H, Maria Bordin da Silva Chacur N, Dias Alves D, Cadore Mafaldo R, Dias Gomes L, Dos Santos Barreto G. Gluteal Augmentation with Polymethyl Methacrylate: A 10-year Cohort Study. Plast Reconstr Surg Glob Open. 2019 May 31;7(5):e2193. doi: 10.1097/GOX.0000000000002193. eCollection 2019 May. PMID 31333932
- [Background] Serra MS, Goncalves LZ, Ramos-e-Silva M. Soft tissue augmentation with PMMA-microspheres for the treatment of HIV-associated buttock lipodystrophy. Int J STD AIDS. 2015 Mar;26(4):279-84. doi: 10.1177/0956462414536878. Epub 2014 May 22. PMID 24855130
- [Background] Atiyeh B, Ghieh F, Oneisi A. Safety and Efficiency of Minimally Invasive Buttock Augmentation: A Review. Aesthetic Plast Surg. 2023 Feb;47(1):245-259. doi: 10.1007/s00266-022-03049-5. Epub 2022 Aug 23. PMID 35999464
- [Background] Dai Y, Chen Y, Hu Y, Zhang L. Current Knowledge and Future Perspectives of Buttock Augmentation: A Bibliometric Analysis from 1999 to 2021. Aesthetic Plast Surg. 2023 Jun;47(3):1091-1103. doi: 10.1007/s00266-022-03140-x. Epub 2022 Oct 25. PMID 36284000
- [Background] de Melo Carpaneda E, Carpaneda CA. Adverse results with PMMA fillers. Aesthetic Plast Surg. 2012 Aug;36(4):955-63. doi: 10.1007/s00266-012-9871-8. Epub 2012 Mar 22. PMID 22437333
- [Background] Ridwan-Pramana A, Idema S, Te Slaa S, Verver F, Wolff J, Forouzanfar T, Peerdeman S. Polymethyl Methacrylate in Patient-Specific Implants: Description of a New Three-Dimension Technique. J Craniofac Surg. 2019 Mar/Apr;30(2):408-411. doi: 10.1097/SCS.0000000000005148. PMID 30676441
- [Background] Carvalho Costa IM, Salaro CP, Costa MC. Polymethylmethacrylate facial implant: a successful personal experience in Brazil for more than 9 years. Dermatol Surg. 2009 Aug;35(8):1221-7. doi: 10.1111/j.1524-4725.2009.01216.x. Epub 2009 May 12. PMID 19438669
- [Background] de la Guardia C, Virno A, Musumeci M, Bernardin A, Silberberg MB. Rheologic and Physicochemical Characteristics of Hyaluronic Acid Fillers: Overview and Relationship to Product Performance. Facial Plast Surg. 2022 Apr;38(2):116-123. doi: 10.1055/s-0041-1741560. Epub 2022 Feb 3. PMID 35114708
- [Background] Clark DP, Hanke CW, Swanson NA. Dermal implants: safety of products injected for soft tissue augmentation. J Am Acad Dermatol. 1989 Nov;21(5 Pt 1):992-8. doi: 10.1016/s0190-9622(89)70288-7. PMID 2681290
- [Background] Jordan DR. Soft-tissue fillers for wrinkles, folds and volume augmentation. Can J Ophthalmol. 2003 Jun;38(4):285-8. doi: 10.1016/s0008-4182(03)80093-5. PMID 12870861
- [Background] Haneke E. Polymethyl methacrylate microspheres in collagen. Semin Cutan Med Surg. 2004 Dec;23(4):227-32. doi: 10.1016/j.sder.2004.08.002. PMID 15745230
- [Background] Blanco Souza TA, Colome LM, Bender EA, Lemperle G. Brazilian Consensus Recommendation on the Use of Polymethylmethacrylate Filler in Facial and Corporal Aesthetics. Aesthetic Plast Surg. 2018 Oct;42(5):1244-1251. doi: 10.1007/s00266-018-1167-1. Epub 2018 Jun 5. PMID 29872906